CLINICAL TRIAL: NCT01137487
Title: Impact of Not Measuring Residual Gastric Volume on Nosocomial Pneumonia Rates in Mechanically Ventilated Patients Receiving Early Enteral Feeding: a Randomized-controlled Study
Brief Title: Study of Impact of Not Measuring Residual Gastric Volume on Nosocomial Pneumonia Rates
Acronym: NUTRIREA1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUTRIREA1
Record Dates: First submitted 2010-05-19; First posted 2010-06-04 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Ventilation-Associated Pneumonia
Keywords: mechanical ventilation; enteral nutrition; Ventilation-Associated Pneumonia; residual gastric volume measurement; vomiting; gastro-oesophageal reflux; early enteral nutrition; Intensive care unit; Enteral Feeding
MeSH Terms: conditions — Vomiting; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- residual gastric volume (Other)
  Interventions: Procedure: monitoring of residual gastric volume
- residual gastric volume not monitored (Other)
  Interventions: Procedure: not monitoring of residual gastric volume

INTERVENTIONS:
Procedure: monitoring of residual gastric volume — measurements of residual gastric volume every six hours in patients receiving early enteral feeding and mechanical ventilation
  Other Names: Residual Gastric Volume Measurement
  Arms: residual gastric volume
Procedure: not monitoring of residual gastric volume — no measurements of residual gastric volume
  Other Names: Non residual Gastric Measurement
  Arms: residual gastric volume not monitored

SUMMARY:
Early enteral feeding is a key component of the management of critically ill patients receiving mechanical ventilation. However, enteral feeding has been associated with serious complications such as aspiration followed by ventilator-associated pneumonia (VAP). Many critically ill patients experience poor tolerance of early enteral nutrition because of impaired gastric motility, which leads to a sequence of delayed gastric emptying, increased gastric volume, gastroesophageal reflux, vomiting, aspiration, and VAP. Routine monitoring of residual gastric volume (RGV) to minimize the risk of aspiration is standard practice. RGV is assumed to reflect gastric content, with high RGVs indicating impaired gastric emptying that requires discontinuation of enteral feeding in order to prevent aspiration.However, RGV measurement is neither standardized nor validated. The cut-off value that may indicate an increased risk of aspiration and therefore a need for discontinuing enteral feeding has not been determined, and cut-offs used in studies have ranged from 150 to 500 ml. No data are available to support a correlation between RGV and the rates of adverse events. In experimental studies, RGV failed to correlate with vomiting, aspiration, or VAP. The investigators hypothesize that RGV monitoring fails to decrease the risk of VAP and leed to inappropriate interruptions in enteral feeding with a risk of underfeeding. To assess the effects of not measuring RGV on VAP and enteral feeding delivery, the investigators designed a prospective randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with invasive mechanical ventilation
* Feeding via nasogastric tube within 36 hours after the initiation of endotracheal mechanical ventilation.
* Age over 18 years
* Informed consent

Exclusion Criteria:

* Mechanical ventilation started more than 36 hours before institution of enteral feeding
* Patients turned in the prone position at inclusion
* Abdominal surgery within 1 month before inclusion
* History of esophageal or gastric surgery
* EN via a gastrostomy or a jejunostomy
* Bleeding from esophagus, stomach or bowel
* Moribund patient
* Age less than 18 years
* Pregnancy.
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To compare ventilator associated pneumonia rates in patients receiving early enteral feeding without residual gastric volume (RGV) monitoring and in patients with RGV monitoring | until weaning of mechanical ventilation (average : 14 days)

SECONDARY OUTCOMES:
mortality rate | 60 days
vomiting rates | until weaning of mechanical ventilation (average : 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, MD, PhD, Principal Investigator — CHD Vendée
Locations (6):
- France (6):
  - CH Angoulème - Réanimation Polyvalente, Angoulême
  - CHD Vendée - Service de Réanimation, La Roche-sur-Yon
  - CHU Limoges - Réanimation Polyvalente, Limoges
  - CHU Orléans - Réanimation Médicale, Orléans
  - CHU Poitier - Réanimation Médicale, Poitiers
  - CHU Tours - Réanimation Polyvalente, Tours

REFERENCES:
- [Derived] Reignier J, Mercier E, Le Gouge A, Boulain T, Desachy A, Bellec F, Clavel M, Frat JP, Plantefeve G, Quenot JP, Lascarrou JB; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Effect of not monitoring residual gastric volume on risk of ventilator-associated pneumonia in adults receiving mechanical ventilation and early enteral feeding: a randomized controlled trial. JAMA. 2013 Jan 16;309(3):249-56. doi: 10.1001/jama.2012.196377. PMID 23321763